CLINICAL TRIAL: NCT02247752
Title: Follow-up of HBsAg Inactive Carriers Study
Acronym: PIBAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Collaborators: INSERM U785-CNR Hôpital Paul Brousse 94800 VILLEJUIF (Unknown); Faculté de mathématiques ORLEANS (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHRO -2014-02
Record Dates: First submitted 2014-09-15; First posted 2014-09-25 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Hepatitis B
Keywords: hepatitis; HBV; chronic hepatitis; HCC; cirrhosis; quantitative HBsAg; HBsAg inactive carriers
MeSH Terms: conditions — Hepatitis B; Hepatitis; Hepatitis, Chronic; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inactive carriers (Other)
  Interventions: Other: inactive carrier

INTERVENTIONS:
Other: inactive carrier — Yearly demographic, clinic, biologic and ultrasonic data collection realized during usual follow-up as recommended.
  Yearly centralisation of a complementary biological analysis in Paul Brousse Hospital laboratory of virology.

SUMMARY:
The definition of HBs antigen (HBsAg) inactive carrier status has evolved during time. We spoke first from HBsAg" healthy carrier ", then from " asymptomatic carrier ", last from HBsAg" inactive carrier ". This definition continue to be not totally consensual. A very low viral load (< 2000 UI/ml) or undetectable, associated with repetitive normal transaminases and with detectable anti-HBe antibodies were necessary to affirm the inactive carrier status on 2009 EASL recommendations. The 2012 EASL recommendations confirm that the normality of alanine aminotransferase (ALT) with an upper limit of normal (ULN) approximately below 40 UI/ml, like low viral load (HBV-DNA), does necessary be verified every 3 or 4 months during a year to diagnose an inactive carrier. Nevertheless, they admit the possibility for some patients to be inactive carriers with HBV-DNA between 2000 and 20000 UI/ml with consistently normal transaminases This study will follow-up HBsAg inactive carriers during 5 years, in order to evaluate the incidence of unfavourable liver events: chronic hepatits B, liver cirrhosis, hepatocarcinoma (CHC) during this time, and to determine the independant prognosis criteria of unexpected arrival of such events. Secondary outcomes will evaluate HBsAg quantification for the prognosis of such events or, in contrary HBs seroconversion; will evaluate the influence of B genotype on HBsAg level; will evaluate the influence of comorbidities on unexpected arrival of such events.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg + since one year or more.

  * HBeAg -, anti-HBe antibodies +
  * HBV-DNA < 20000 UI/ml on all dosages realized during past year (ultra-sensitive PCR with a detection threshold < 20 UI/ml), at least 2 dosages during past year.
  * AST and ALT transaminases < ULN on all dosages realized during past year (at least 3).
  * Age > 18 and < 70
  * We will include consecutively all encountered patients (consultation, hospitalization) and diagnosed as HBsAg inactive carriers in each participating center.

Exclusion Criteria:

* anti-VHC antibodies +
* anti-VHD antibodies +
* anti-VIH antibodies +
* genetic hemochromatosis
* liver cirrhosis on liver biopsy or with non-invasive methods (Fibrometer, Fibroscan, Fibrotest, Hepascore …)
* Past or present treatment against HBV
* Ultrasonic diagnosis of HCC or Portal Hypertension
* non compliant patient whom 5 years follow-up seems uncertain.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 619 (Actual)
Dates: Start 2014-09-16 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Incidence of unfavourable liver events | every year, during 5 years for each
  The primary outcome that the study was designed to evaluate is the incidence of unfavourable liver events (chronic hepatitis B, liver cirrhosis, HCC) in a cohort of patients presumed to be " HBsAg inactive carriers ".

CONTACTS AND LOCATIONS:
Overall Officials: Xavier CAUSSE, Principal Investigator — CHR Orleans
Locations (32):
- France (32):
  - Ch General Du Pays D'Aix, Aix-en-Provence
  - CH d'AVIGNON, Avignon
  - Clinique de La Chataigneraie, Beaumont
  - Medical Center Besancon, Besançon
  - Clinical Center Bourgoin Jallieu, Bourgoin
  - Hopital Sainte Camille, Bry-sur-Marne
  - Ch de Caen, Caen
  - Ch Sud Fracilien Jean Jaures, Corbeil-Essonnes
  - CH CREIL, Creil
  - Ch de Creteil, Créteil
  - CH de GONESSE, Gonesse
  - Clinique Du Palais, Grasse
  - Ch D'Hyeres, Hyères
  - Ch de Lagny Marne La Valee, Jossigny
  - Chd Vendee, La Roche-sur-Yon
  - Ch Du Mans, Le Mans
  - Medical Center La Sauvegarde, Lyon
  - Ch de Meaux, Meaux
  - CH MELUN, Melun
  - Ch Montelimar, Montélimar
  - Ch de Montfermeil, Montfermeil
  - Clinical Center Montpellier, Montpellier
  - Medical Center Nanterre, Nanterre
  - CHR d'ORLEANS, Orléans
  - Medical Center Paris 7, Paris
  - Ch de Pau, Pau
  - Hopital Saint Jean, Perpignan
  - Ch de La Region Annnecienne, Pringy
  - Ch Saint Brieuc, Saint-Brieuc
  - Ch de Saint Denis, Saint-Denis
  - Ch de Vannes, Vannes
  - Chi Villeneauve Saint Georges, Villeneuve-Saint-Georges